CLINICAL TRIAL: NCT05063864
Title: Determining the Effectiveness of the Post-Hysterectomy Nursing Support Program: Randomized Controlled Study
Brief Title: Post-Hysterectomy Nursing Support Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Kübra Yılmaz, Principal Investigator, Suleyman Demirel University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KYilmaz
Record Dates: First submitted 2021-09-01; First posted 2021-10-01 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Hysterectomy
Keywords: hysterectomy; nursing support program,; menopausal symptoms; sexuality; depression; quality of life
MeSH Terms: conditions — Sexuality; Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nursing Support Program (Experimental): the group that applied the nursing support program
  Interventions: Other: Nursing Support Program
- No Nursing Support Program (No Intervention): the group that did not receive a nursing support program

INTERVENTIONS:
Other: Nursing Support Program — Within the scope of the nursing support program, counselling services were provided to women by making regular phone calls that lasted 15-20 minutes once a week. Within the scope of the support program, two training booklets titled "Life After Hysterectomy Surgery" and "Women's Health During Menopause" were prepared by reviewing the literature.
  Arms: Nursing Support Program

SUMMARY:
Objective: This study was conducted to evaluate the effectiveness of the nursing support program developed for women undergoing hysterectomy.

Background: Hysterectomy is an important surgical intervention that affects women physically, sexually and psychosocially.

Method: The study is a single blind, randomized controlled study conducted at the Department of Obstetrics and Gynecology in a university hospital between November 2017 and November 2018. 60 women who had hysterectomy were divided into experimental and control groups and It was evaluated on the 1-2 day, 6-7 day and 2nd month. In the study, the nursing support program was applied only to women in the experimental group.

DETAILED DESCRIPTION:
Aim: This study was conducted to evaluate the effectiveness of the nursing support program developed for women who had hysterectomy.

Methods: A prospective, randomised controlled study was conducted in the gynaecology clinic of a university hospital between November 2017 and November 2018. It was conducted in a single-blind, randomised controlled trial with a total of 60 women in the experimental and control groups. A nursing support program had been developed for women who have had a hysterectomy. The program developed for the experimental group and the routine program for routine maintenance and control group were applied. The initial evaluation was carried out postoperative on the 1st-2nd day, the second assessment was carried out on the 6th-7th day and the third evaluation was carried out at 2 months. The first interview was carried out in the hospital, and the second and third interviews were carried out with home visits. The sociodemographic data form, postoperative evaluation form, Female Sexual Function Index (FSFI), Epidemiological Studies and Central Depression Scale (EAMDS), Menopausal Symptoms Evaluation Scale (MSDS) and SF-12 quality of life scale were used to collect data.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis benign hysterectomy and bilateral oophorectomy
* Having no communication problems.

Exclusion Criteria:

* Clinical diagnosis vaginal hysterectomy
* Clinical diagnosis psychiatric disorders and therefore used drugs

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2019-06-24 (Actual)

PRIMARY OUTCOMES:
Nursing Support Program | postoperative on the 2 months.
  Change of postoperative symptoms in the postoperative data sheet at 2 months after hysterectomy, Change of sexual functions in female sexual function index (FSFI) 2 months after hysterectomy Change of mental status in epidemiological depression scale (CES-D) 2 months after hysterectomy Change in quality of life in SF-12 quality of life scale at 2 months after hysterectomy Change in menopausal symptoms in the menopausal symptoms rating scale (MRS) 2 months after hysterectomy

CONTACTS AND LOCATIONS:
Overall Officials: Kübra Yilmaz, Principal Investigator — Suleyman Demirel University
Locations (1):
- Suleyman Demirel University, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I am not sure.